CLINICAL TRIAL: NCT00578045
Title: UARK 2006-28 Human Cord Blood Transplantation in Advanced Hematological Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no accrual
Sponsor: University of Arkansas (Other)
Responsible Party: Frits van Rhee, MD, PhD, University of Arkansas for Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 67363
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Approximately 24 hours after the chemotherapy is completed you will receive the transfusion of the human cord blood
  Interventions: Procedure: Transfusion

INTERVENTIONS:
Procedure: Transfusion — Approximately 24 hours after the chemotherapy is completed you will receive the transfusion of the human cord blood

SUMMARY:
The researchers want to find out if subjects treated on this study will achieve long term bone marrow recovery (engraftment) and if their tumors will respond to this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced hematological malignancies who have failed at least two lines of therapy.
* Karnofsky performance score > 60, unless due to disease and then > 50.
* Age > 18 years.
* An expected survival of > 3 months.
* Subjects must have signed an IRB-approved consent and been informed about the investigational nature of the study.
* Cord blood must have negative serology for HIV.
* Release of cord blood.
* The nucleated cell count of the CBU shall equal or exceed 1 x 107 per kg of recipient body weight.

Exclusion Criteria:

* Liver function: total bilirubin > 2x ULN or AST/ALT > 3x ULN.
* Creatinine > 3.0 mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The researchers on this study want to find out if subjects treated on this study will achieve long term bone marrow recovery (engraftment) and if their tumors will respond to this treatment. | 12 months

SECONDARY OUTCOMES:
The researchers also want to find out what types of side effects, if any, subjects will experience with this treatment. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States